CLINICAL TRIAL: NCT05769452
Title: Effect of Closed Intravenous Catheter System on Catheter Success, Length of Stay and Complications in Pediatric Hematology and Oncology Patients
Brief Title: Closed Intravenous Catheter System on Catheter Success, Length of Stay and Complications
Acronym: nexiva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gülçin Özalp Gerçeker (Other)
Responsible Party: Sponsor-Investigator, Gülçin Özalp Gerçeker, pHD, Assoc. Prof., Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DEU PHO nexiva
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Catheter Complications; Catheter Leakage
Keywords: closed IV catheter system; pediatric hematology oncology; first IV attempt

STUDY DESIGN:
Intervention Model Description: In this study, the intervention group was given a closed IV catheter system called BD Nexiva™; the control group received an open IV catheter called BD Insyte™ Autoguard™. Within the scope of the study, "Peripheral IV Catheter Care Bundle Approach" was applied to all patients.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BD Nexiva™ (Experimental): The intervention group was given a closed IV catheter system called BD Nexiva™.
  Interventions: Device: closed IV catheter system (BD Nexiva™)
- BD Insyte™ Autoguard™ (Experimental): The control group received an open IV catheter called BD Insyte™ Autoguard™.
  Interventions: Device: open IV catheter (BD Insyte™ Autoguard™)

INTERVENTIONS:
Device: closed IV catheter system (BD Nexiva™) — There is a high-pressure extension set and a Q-syte split septum needle-free intervention device at the tip of the catheter. It creates a closed integrated system with this apparatus, reducing the risk of catheter-related bloodstream infection.
  Other Names: BD Nexiva™
  Arms: BD Nexiva™
Device: open IV catheter (BD Insyte™ Autoguard™) — BD Instaflash™ needle technology improves initial entry success by confirming vascular access through the needle noch. It has flexible wings for secure cannula fixation.
  Other Names: BD Insyte™ Autoguard™
  Arms: BD Insyte™ Autoguard™

SUMMARY:
Peripheral intravenous catheters (PIVCs) can be used frequently in pediatric hematology oncology patients. There are different types of PIVCs as open and closed. There are studies on adults using the closed IV catheter system, which is a type of PICK. However, no study was found in the literature in which the closed IV catheter system was used in the pediatric population.

DETAILED DESCRIPTION:
The primary purpose of this research is; to evaluate the effect of two different catheter systems (closed IV catheter system: BD Nexiva™/ peripheral open IV catheter: BD Insyte™ Autoguard™) on catheter stay in pediatric hematology and oncology patients aged 1-12 years.

The secondary aim of the research is; to evaluate the effect of two different catheter systems on the success of catheter placement and the development of complications in the first attempt in pediatric hematology and oncology patients.

ELIGIBILITY:
Inclusion Criteria:

* Age range of pediatric patients is between 1-12
* Obtaining an informed consent form from the child patient and parent
* Child patient receiving intravenous therapy

Exclusion Criteria:

* port or central venous catheter in the pediatric patient

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
catheter indwelling time | during the catheterization
  time between catheter insertion and removal
success of catheter placement | at catheter insertion
  first IV attempt

SECONDARY OUTCOMES:
development of catheter complications | during the catheterization
  infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Nur Olgun, MD, Principal Investigator — Dokuz Eylul University; Hale Ören, MD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozalp Gerceker G, Yildirim BG, Onal A, Oren H, Olgun HN, Bektas M. The effect of the closed intravenous catheter system on first insertion success, indwelling time, and complications in pediatric hematology and oncology patients: A randomized controlled study. Eur J Oncol Nurs. 2023 Dec;67:102430. doi: 10.1016/j.ejon.2023.102430. Epub 2023 Oct 7. PMID 37879193